CLINICAL TRIAL: NCT07098520
Title: Biomarkers of Steatohepatitis in Type 2 Diabetes Patients
Acronym: STEDIB
Status: Not yet recruiting | Type: Observational
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Jan Polak, physician, principal investigator, Faculty Hospital Kralovske Vinohrady
Other Study IDs: STEDIB
Record Dates: First submitted 2024-04-27; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Diabetes; Steatosis of Liver
MeSH Terms: conditions — Diabetes Mellitus; Fatty Liver

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and serum aliquots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diabetes type 2: Patients diagnosed with type 2 diabetes
  Interventions: Other: No intervention, just observation

INTERVENTIONS:
Other: No intervention, just observation — no intervention, study investigates biomarkers associated with a disease

SUMMARY:
The aims of the study are to identify a subgroup of type 2 diabetics at risk of developing and progressing to non-alcoholic steatohepatitis (NASH), to correlate clinical and laboratory parameters with sonographic and elastographic findings in order to pinpoint indicators of liver fibrosis (NASH), and to facilitate targeted screening and intensified management of type 2 diabetes mellitus to prevent NASH complications.

DETAILED DESCRIPTION:
Hepatic steatosis, known as non-alcoholic fatty liver disease (NAFLD), is prevalent among type 2 diabetes mellitus patients. NAFLD encompasses benign hepatic steatosis and non-alcoholic steatohepatitis (NASH), the latter being a hepatic complication linked to metabolic syndrome. Insulin resistance and dysregulation of fatty acid metabolism contribute to its pathogenesis, leading to oxidative stress, hepatocyte damage, and fibroproduction, eventually progressing to cirrhosis and hepatocellular carcinoma.

Identification of high-risk NAFLD patients, particularly those with NASH, is crucial for early intervention and monitoring. However, distinguishing between benign steatosis and NASH poses a clinical challenge. Liver biopsy remains the gold standard for NASH diagnosis but is invasive and impractical for routine screening in diabetic patients.

The study aims to identify high-risk type 2 diabetics prone to NASH progression by correlating clinical and laboratory parameters with sonographic and elastographic findings. Parameters such as diabetes duration, BMI, waist/hip ratio, glycated hemoglobin, and liver function tests will be compared with real-time shear wave elastography results. This approach seeks to pinpoint indicators of liver fibrosis (NASH), facilitating targeted screening and intensified management of type 2 diabetes mellitus, potentially averting NASH complications.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes diagnosis

Exclusion Criteria:

Alcohol abuse (anamnestic) Hepatitis Other known liver disease (other than steatosis/steatohepatitis)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with Type 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
FIB-4 (Fibrosis-4) index | Cross sectional study - one day of clinical investigation
  FIB-4 index - marker of liver fibrosis (calculated from variables provided below) will be evaluated in all subjects.
  FIB-4 index is calculated as follows: FIB-4 = (Age × AST) / (Platelets × √ALT). This requires values: the patient's age in years, AST (aspartate aminotransferase) in U/L, ALT (alanine aminotransferase) in U/L, and platelet count in 10^9/L.
  A score below 1.3 suggests minimal fibrosis, while a score above 3.25 indicates advanced fibrosis.

SECONDARY OUTCOMES:
ELF (Enhanced Liver Fibrosis) score | Cross sectional study - one day of clinical investigation
  ELF (Enhanced Liver Fibrosis) score will be determined in all subjects.
  The ELF score is calculated as follows: ELF score = 2.278 + 0.851 × ln(HA) + 0.751 × ln(PIIINP) + 0.394 × ln(TIMP-1), where HA represents serum concentration of hyaluronic acid in ng/mL, PIINP represents serum concentration of procollagen III N-terminal peptide in ng/mL and TIMP-1 represents serum concentration of tissue inhibitor of metalloproteinase in ng/mL.
  The reference range of the ELF score (7.14-9.55), higher values suggest more advanced liver fibrosis.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study will be provided to qualified researchers with a legitimate research interest.
Supporting Information: Study Protocol
Time Frame: The data will be made available starting 6 months after the study completion date for 10 years.
Access Criteria: Access to the data will be granted following the review and approval of a research proposal and a signed Data Sharing Agreement (DSA). Requests for access can be submitted via email to jan.polak@lf3.cuni.cz